CLINICAL TRIAL: NCT05448131
Title: Towards an Individually Tailored Enzyme Replacement Therapy in Pompe Disease: A Controlled Study for Elucidation of Molecular Structures Contributing to Enzyme Uptake and Immunoreactivity
Brief Title: ERT in Pompe Disease: Elucidation of Molecular Structures Contributing to Enzyme Uptake and Immunoreactivity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre for Analytical Biochemistry and Biomedical Mass Spectrometry (Other)
Collaborators: University of Giessen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Michael Przybylski, Professor of Analytical Biochemistry, Centre for Analytical Biochemistry and Biomedical Mass Spectrometry
Other Study IDs: SGZ-2020-13329
Record Dates: First submitted 2022-06-29; First posted 2022-07-07 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Pompe-Disease
Keywords: Antibodies
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
In the first part of this study, the aim is to characterize the molecular structure of wildtype GAA and, in particular, of mutated GAA variants with and without HSAT, in order to learn how mutation impairs uptake of GAA into the cell via the M6P receptor. In the second part of the study the aim is to learn to which epitopes antibodies bind and to which not. To accomplish this the investigators will synthesize and chemically modify the epitope peptides, in order to block effectively antibodies directed against the therapeutic enzyme.

DETAILED DESCRIPTION:
Enzyme replacement therapy (ERT) with recombinant human GAA (rhGAA = alglucosidase alfa) is available since 2006, and has been shown effective in IOPD and LOPD; however the treatment response is variable and imperfect. This has prompted the development of a next-generation rhGAA with increased glycosylation and improved muscle cell uptake (avalglucosidase alfa). The efficacy of ERT significantly depends on the glycosylation status of the enzyme determining muscle cell uptake via the mannose-6-phosphate (M6P) receptor, and on the formation of antibodies directed against the recombinant enzyme. The impact of immunological factors on efficacy is highlighted by the occurrence of high sustained antibody titers (HSAT) in IOPD patients producing no GAA at all (CRIM-negative), that result in a worse outcome similar to that of untreated patients, if no immunomodulating medication is given. Such HSAT can also occur in IOPD patients synthesizing a non-functional GAA (CRIM-positive) and in some late onset Pompe Disease (LOPD) patients.

In the first part of this study, the investigators aim to characterize the molecular structure of wildtype GAA and, in particular, of mutated GAA variants with and without HSAT, in order to learn how mutation impairs uptake of GAA into the cell via the M6P receptor. To accomplish this, 5 healthy subjects and 45 Pompe disease patients will be studied (15 IOPD and 30 LOPD). The investigators will identify antibody epitopes in the sera of patients with rhGAA antibodies and determine and compare quantitatively their binding affinities, by using a combination of proteolytic affinity-mass spectrometry and surface plasmon resonance biosensor analysis. The investigators reason that specific mutations may affect the epitope status differently. Related to this, the investigators also speculate that glycosylations and M6P residues could modify epitopes in their close vicinity. These results will help to understand where the antibody binding epitopes are located.

In the second part of the study the investigators aim to learn to which epitopes antibodies bind and to which not. To accomplish this the epitope peptides will be synthesized and chemically modified, in order to block effectively antibodies directed against the therapeutic enzyme. Applying high affinity GAA epitope peptides capable of binding neutralizing antibodies is expected to potentially improve efficacy and safety of ERT, thereby providing a new targeted and personalized immunotolerance approach.

ELIGIBILITY:
Inclusion Criteria:

* All patients or their legal guardian and healthy volunteers with normal GAA enzyme activity and genotype will give informed consent to participate in this explorative, cross-sectional study.
* IOPD/LOPD patients will have a confirmed diagnosis of Pompe disease based on enzyme activity reduction and genetic GAA mutations.
* Both CRIM-positive and CRIM-negative IOPD patients will be included.
* Patients with IOPD/LOPD will be on enzyme replacement therapy on their individual treatment regime.
* Healthy volunteers will be included as controls for wildtype GAA analysis.

Exclusion Criteria:

* Patient/healthy volunteer or legal guardian do not agree to give informed consent.
* The patient/healthy volunteer is not capable to adhere to the study protocol.
* The patient is not treated with enzyme replacement therapy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 50 patients who meet all eligibility criteria will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-08-06 (Estimated); Study Completion 2024-10-07 (Estimated)

PRIMARY OUTCOMES:
Determination of epitope numbers of acid-alpha-glucosidase (wtGAA; rhGAA; mutated GAA) antibodies | Only at baseline visit
  Epitope numbers of wtGAA, rhGAA, and mutated GAAs will determine the number of Pompe patients with polyclonal and monoclonal antibodies, and determine whether specific antibodies are more prevalent than others among Pompe patients.
Determination of epitope locations of acid-alpha-glucosidase (wtGAA; rhGAA; mutated GAA) antibodies | Only at baseline visit
  Epitope locations of wtGAA, rhGAA, and mutated GAAs will determine the number of Pompe patients with polyclonal and monoclonal antibodies, and determine whether specific antibody epitopes are more prevalent than others among Pompe patients.
Determination of epitope- specific affinities of acid-alpha-glucosidase (wtGAA; rhGAA; mutated GAA) antibodies | Only at baseline visit
  Epitope- specific affinities of acid-alpha-glucosidase (wtGAA; rhGAA; mutated GAA) antibodies in PD patients will be determined for correlation with mutations in GAA structure

SECONDARY OUTCOMES:
Determination of the number of PD patients with specific neutralizing antibody epitopes | Only at baseline visit
  Neutralizing antibodies in PD patients may be differentiated by their epitope specificities.
Determination of antibody titers in PD patients | Only at baseline visit
  Determination of epitope-specific antibody titers

OTHER OUTCOMES:
Identification of the feasibility of epitope peptides for molecular apheresis of antibodies. | Only at baseline visit
  Quantitative determination of binding capacity of identified epitope peptides of PD patients to enable molecular apheresis of antibodies.
  To compare the antibody/epitope data obtained in this study with IARs and GAA antibody classes determined in the Sanofi-Genzyme lab.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Przybylski, PhD, Principal Investigator — Centre for Analytical Biochemistry, 65428 Ruesselsheim am Main, Germany
Locations (1):
- Centre for Analytical Biochemistry, Rüsselsheim am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No